CLINICAL TRIAL: NCT03615742
Title: Diesel Exhaust Induces Glucocorticoid Resistance
Acronym: DIGR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); AllerGen NCE Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Carlsten, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: H17-01336
Record Dates: First submitted 2018-07-23; First posted 2018-08-06 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Exposure to Pollution; Glucocorticoid Resistance
Keywords: Diesel Exhaust; Air Pollution; Inhaled Corticosteroids; Gene Expression; Asthma; Controlled Human Exposure Study
MeSH Terms: conditions — Glucocorticoid Receptor Deficiency; Asthma | interventions — Budesonide; Vehicle Emissions

STUDY DESIGN:
Intervention Model Description: Volunteers will visit our lab four different times to be exposed to: 1) placebo & filtered air, 2) placebo & diesel exhaust, 3) budesonide and filtered air, and 4) budesonide and diesel exhaust
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding of exposures will be performed by the air pollution exposure laboratory (APEL) engineer, who will not interact with volunteers. Visually indistinguishable placebo and budesonide inhalers will be coded by research pharmacy staff. All assays will be performed by personnel who do not know the exposure conditions of individual samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo and Filtered Air (Placebo Comparator): Volunteers will use an inhaler that does not contain any medication, before sitting in a booth and being exposed to high-efficiency particulate air (HEPA) filtered air for 2 hours.
  Interventions: Other: Placebo; Other: Filtered Air
- Budesonide and Filtered Air (Active Comparator): Volunteers will inhale 1.6mg of budesonide before sitting in a booth and being exposed to HEPA filtered air for 2 hours.
  Interventions: Drug: Budesonide; Other: Filtered Air
- Placebo and Diesel Exhaust (Active Comparator): Volunteers will use an inhaler that does not contain any medication, before sitting in a booth and being exposed to 300µg/m³ concentration of diesel exhaust for 2 hours.
  Interventions: Other: Placebo; Other: Diesel Exhaust
- Budesonide and Diesel Exhaust (Experimental): Volunteers will inhale 1.6mg of budesonide before sitting in a booth and being exposed to 300µg/m³ concentration of diesel exhaust for 2 hours.
  Interventions: Drug: Budesonide; Other: Diesel Exhaust

INTERVENTIONS:
Other: Placebo — Inhalation of air through a Turbuhaler that contains no medication, as a control.
  Arms: Placebo and Diesel Exhaust; Placebo and Filtered Air
Drug: Budesonide — 1.6mg of budesonide from a Turbuhaler.
  Other Names: Pulmicort
  Arms: Budesonide and Diesel Exhaust; Budesonide and Filtered Air
Other: Filtered Air — Exposure to HEPA filtered air, as a control.
  Arms: Budesonide and Filtered Air; Placebo and Filtered Air
Other: Diesel Exhaust — Diesel exhaust standardized to 300µg/m³ of particulate matter with a diameter of 2.5 micrometers or less (PM2.5).
  Other Names: Traffic Related Air Pollution
  Arms: Budesonide and Diesel Exhaust; Placebo and Diesel Exhaust

SUMMARY:
The investigators are studying the effects of exposure to diesel exhaust on lung inflammation in the presence and absence of an inhaled corticosteroid. Although data is mixed, studies show that asthmatics have increased lung inflammation and worse symptoms during periods of higher air pollution despite taking their anti-inflammatory corticosteroid medication. One possible reason is that air pollution exposure may decrease the ability of corticosteroids to combat inflammation.

To test this volunteers will inhale either a placebo or a corticosteroid, before sitting in an exposure booth for 2 hours breathing either filtered air or diluted diesel exhaust. Samples will be collected before and after exposure to analyze the effects of budesonide and diesel exhaust exposure.

DETAILED DESCRIPTION:
1) Purpose Inhalation of air pollutants leads to both airway inflammation, with increased cytokine expression and inflammatory cell recruitment to the airways, and to airway hyperresponsiveness, which together contribute to airway resistance and breathing difficulties. Correlational data indicate that exposure to air pollution increases inhaled corticosteroids (ICS) use in asthmatics, suggesting that steroidal anti-inflammatory medications are suboptimally effective under these conditions. However, a major issue is that no study has yet been performed specifically to determine the effects of controlled diesel exhaust (DE) exposure on responses to ICS. Furthermore, investigators need better insight into mechanisms, including the effects of epigenetic modifications and polymorphisms in oxidative stress response genes, which remain under explored. Investigators anticipate that an improved understanding of air pollution-induced ICS hyporesponsiveness (reduced effectiveness) could underpin preventative guidelines, guide ICS usage in response to environmental exposures, and inform rational pharmaceutical development. Ultimately this could lead to fewer exacerbations in asthmatic and other susceptible populations.

Hypothesis:

Acute exposure to DE reduces ICS-inducible gene expression in vivo in asthmatics, in part through effects on epigenetic processes.

Justification:

Air pollution exposure correlates with increased use of ICS inhalers in asthmatics, suggesting that ICS offer less control during periods of higher air pollution. As genes induced by ICS are critical in reducing inflammatory messenger ribonucleic acid (mRNA) and protein expression, the investigators have chosen to focus on the effects of DE on ICS-inducible gene expression as our primary endpoint.

Research Method:

To test this the effects of air pollution exposure on a corticosteroid, volunteers will inhale either a placebo (inhaler containing no medication) or budesonide (1.6mg), before sitting in our exposure booth for 2 hours breathing either filtered air (as a control) or diluted diesel exhaust (standardized to 300µg/m³ of particulate matter with a diameter of 2.5 micrometers or less).

Volunteers will visit our lab four different times to be exposed to: 1) placebo & filtered air, 2) placebo & diesel exhaust, 3) corticosteroid and filtered air, and 4) corticosteroid and diesel exhaust. Investigators can then compare responses to each of these combinations of exposures.

Investigators will take blood samples before and after volunteers complete each of these exposures to track how they affect the body. Six hours after placebo or budesonide inhalation a research bronchoscopy will be performed during which a very thin flexible tube will be inserted through the mouth and down into lungs to collect samples from each volunteer.

Bronchoalveolar lavage, bronchial washes, bronchial brushes and tissue biopsies will be obtained for analysis of gene expression and epigenetic endpoints. Nasal lavage samples will also be collected to examine responses in the upper airways and blood and urine will be studied to examine systemic responses. Spirometry will be used to assess effects on airway function.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19-49
2. Have physician-diagnosed asthma confirmed by the study physician examination, spirometry, methacholine challenge provocative concentration causing a 20% fall (PC20) of <16 mg/mL, and questionnaires during a screening visit

Exclusion Criteria:

1. Smoking of any kind (0.5 pack-years ever, or any current) or use of vape/vaporizing devices
2. Regular anti-histamine, NSAID, corticosteroid or other controller medication use
3. Pregnancy or breastfeeding
4. Methacholine PC20 >16
5. Relevant cardiac condition or arrhythmia
6. Body mass index of >35
7. Currently participating in another study that may interfere with this study
8. Use of either inhaled or oral corticosteroids in preceding 6 months
9. Substantial comorbidities on study physician's examination or other concerns
10. Surgery scheduled before anticipated study completion

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in DNA methylation, mRNA and protein expression attributable to diesel exhaust and inhaled corticosteroid | Baseline versus 6 hours
  EPIC arrays and RNA Seq will be used to determine effect of exposure(s)

SECONDARY OUTCOMES:
Modification by variants in genes governing inflammation and responses to oxidative stress after DE exposure and ICS. | Baseline versus 6 hours
  Genotypes will be assessed using Applied Biosystems Axiom Precision Medicine Research arrays, with validation by polymerase chain reaction assay (PCR). The data generated will be used to generate a gene score (single value for each participant) which will be used for statistical interaction analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Carlsten, MD, Principal Investigator — University of British Columbia; Christopher F Rider, PhD, Study Director — University of British Columbia; Robert Newton, PhD, Study Director — University of Calgary
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No